CLINICAL TRIAL: NCT03817515
Title: Expanded Access for an Intermediate-size Population for ABI-009 (Sirolimus Albumin-bound Nanoparticles for Injectable Suspension) in Patients With Advanced Perivascular Epithelioid Cell Tumors (PEComa) and Patients With a Malignancy With Relevant Genetic Mutations or mTOR Pathway Activation
Brief Title: Expanded Access for ABI-009 in Patients With Advanced PEComa and Patients With a Malignancy With Relevant Genetic Mutations or mTOR Pathway Activation
Status: Approved for marketing | Type: Expanded Access
Sponsor: Aadi Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PEX-002
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: PEComa, Malignant; TSC1; TSC2; mTOR Pathway Abberation
MeSH Terms: conditions — Perivascular Epithelioid Cell Neoplasms

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: ABI-009 — Sirolimus Albumin-bound Nanoparticles
  Other Names: nab-sirolimus, nab-rapamycin, albumin-bound sirolimus, Sirolimus Albumin-bound Nanoparticles

SUMMARY:
Expanded Access for an Intermediate-size Population for ABI-009 (Sirolimus Albumin-bound Nanoparticles for Injectable Suspension) in Patients with Advanced Perivascular Epithelioid Cell Tumors (PEComa) and Patients with a Malignancy with Relevant Genetic Mutations or mTOR Pathway Activation

DETAILED DESCRIPTION:
Expanded Access for an Intermediate-size Population for ABI-009 (Sirolimus Albumin-bound Nanoparticles for Injectable Suspension) in Patients with Advanced Perivascular Epithelioid Cell Tumors (PEComa) and Patients with a Malignancy with Relevant Genetic Mutations or mTOR Pathway Activation

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for inclusion in this expanded access program only if all of the following criteria are met:

1. a) Diagnosis of advanced (locally advanced and inoperable or metastatic) malignant PEComa confirmed by pathology and immunohistochemistry, whether or not previously exposed to an mTOR inhibitor, or b) diagnosis of any other malignancy with activation in any mTOR pathway component as identified by immunohistochemistry or an identified relevant rare genetic mutation in mTOR pathway genes, including but not limited to TSC1, TSC2, PIK3CA, PTEN, for which there are no FDA-approved treatments or no other comparable or satisfactory alternative therapies available whether or not they been previously exposed to a mTOR inhibitor.
2. 18 years or older, with Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
3. Acceptable blood chemistry levels at screening (obtained ≤14 days prior to enrollment (local laboratory) including:

   1. total bilirubin ≤1.5 x upper limit of normal (ULN)
   2. AST ≤2.5 x ULN (≤5 x ULN if attributable to liver metastases)
   3. serum creatinine ≤1.5 x ULN
4. Adequate biological parameters as demonstrated by the following blood counts at screening (obtained ≤14 days prior to enrollment, local laboratory):

   1. Absolute neutrophil count (ANC) ≥1.5 × 109/L;
   2. Platelet count ≥100,000/mm3 (100 × 109/L);
   3. Hemoglobin ≥8 g/dL.
5. Fasting serum triglyceride <300 mg/dL; fasting serum total cholesterol <350 mg/dL.
6. Male or non-pregnant and non-breast feeding female:

   * Females of child-bearing potential must agree to use effective contraception without interruption from 28 days prior to starting IP and while on investigational medication and have a negative serum pregnancy test (β -hCG) result at screening and agree to ongoing pregnancy testing during the course of the expanded access protocol, and after the end of treatment. A second form of birth control is required even if she has had a tubal ligation.
   * Male patients must practice abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the expanded access protocol. A second form of birth control is required even if he has undergone a successful vasectomy.
7. Ability to understand and sign informed consent.

Exclusion Criteria:

A patient will not be eligible for inclusion in this protocol if any of the following criteria apply:

1. Uncontrolled serious medical or psychiatric illness. Patients with a "currently active" second malignancy other than non-melanoma skin cancers, carcinoma in situ of the cervix, resected incidental prostate cancer (staged pT2 with Gleason Score ≤ 6 and postoperative PSA <0.5 ng/mL), or other adequately treated carcinoma-in-situ are ineligible. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for ≥1 year.
2. In the treating physician's opinion, the potential risks outweigh the potential benefits of therapy with ABI-009.
3. Prior exposure to ABI-009.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult